CLINICAL TRIAL: NCT06541210
Title: Building Community Living Labs (CoLLab) in Black Communities With the Goal of Advancing Prostate Health Equity and Reducing Prostate Cancer Disparities in Black Men
Brief Title: Building Community Living Labs in Black Communities to Advance Prostate Health Equity and Reduce Prostate Cancer Disparities in Black Men
Acronym: CoLLab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-007988; W81XWH-22-PCRP-IDA (Other Grant/Funding Number: Department of Defense); NCI-2024-06410 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CoLLab (Other: Mayo Clinic); 23-007988 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Community Health Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health services research (CoLLab Learning Health System) (Experimental): Participants access CoLLab Learning Health System to use any of the services at least twice monthly for up to 1 year.
  Interventions: Other: Community Health Service; Other: Questionnaire Administration

INTERVENTIONS:
Other: Community Health Service — Access CoLLab Learning Health System to use any of the services
  Other Names: non-interventional study
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial the possibility of establishing a Community Living Labs (CoLLab) Learning Health System to facilitate access to prostate health Risk, Education, and Assessment in the Community with Help (REACH) services in Black men and compares the impact to American Legion Posts with no CoLLab set up at the individual and community levels. Cancer is the second leading cause of death for Black men and Black men are less likely to receive prostate cancer screening. CoLLab Learning Health System utilizes community health workers (CHW) that are well-trained to form a bridge between communities and clinicians. In fact, Black men who work with CHW's typically have better access to health services, gain knowledge about cancer, cancer prevention, treatment and may have better overall health outcomes. Establishing a CoLLab Learning Health System at American Legion Posts may improve access to clinical trials and prostate cancer services in Black men.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Co-create real-life user centric CoLLab Learning Health System at three American Legion Posts, compared to an American Legion Post with no CoLLab set-up. American Legion Post 197 will serve as the hub and Post 244 and Post 194 as the spokes.

II. Assess and evaluate the impact of the CoLLab Learning Health Systems compared to the comparison Post at the individual and community levels.

III. Explore the feasibility of replicating the CoLLab Learning Health System in Black communities nationally.

OUTLINE:

Participants access CoLLab Learning Health System to use any of the services at least twice monthly for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* AIMS 1 AND 3: Participants must be one of the following key personnel:

  * Community PI (n=1),
  * CoLLab Program Manager (n=1)
  * CoLLab Site Managers (n=3)
  * CoLLab CAB members (n=21)
  * 2 Community Health Workers (CHWs) per Post site (n=6)
* AIMS 1 AND 3: Between the ages of 21 and 80.
* AIMS 1 AND 3: Able to complete the survey in English.
* AIMS 1 AND 3: Reside in the Jacksonville, FL and/or surrounding counties.
* AIMS 1 AND 3: Willing and able to consent to the study.
* AIM 2: Black adult of any gender.
* AIM 2: Must be between the ages of 30 and 80.
* AIM 2: Able to speak English.
* AIM 2: Reside in the Jacksonville, FL and/or surrounding counties.
* AIM 2: Willing and able to consent to the study.

Exclusion Criteria:

* AIMS 1 AND 3: Younger than 21years or older than 80 years.
* AIMS 1 AND 3: Not a resident of NE Florida. Unwilling or unable to consent to the study.
* AIM 2: Younger than 30 years or older than 80 years.
* AIM 2: Not a resident of NE Florida.
* AIM 2: Unwilling or unable to consent to the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-05-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Create real-life user centric CoLLab Learning Health System (program production) | Up to 12 months
  Qualitative data collection will be employed during a town hall meeting with the CoLLab Community Advisory Board (CAB) to ensure that we get unbiased and objective feedback from participants.
Impact of the CoLLab Learning Health Systems | Baseline; up to 12 months
  Will be assessed using pre-test and post-test survey scores from a Prostate Health Resources Questionnaire, which consists of 6 multiple choice questions, 8 true/false/don't know questions, 13 questions answered on a 5-point scale (e.g., very favorable to unfavorable or strongly agree to strongly disagree), and 20 yes/no questions.
Feasibility of Replication - cost analysis | Up to 24 months
  Will be assessed using cost analysis of direct and indirect costs.
Feasibility of Replication - qualitative | Up to 24 months
  Will be assessed qualitatively based on interviews of key personnel and users

CONTACTS AND LOCATIONS:
Overall Officials: Folakemi T. Odedina, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials